CLINICAL TRIAL: NCT03242187
Title: (MansTaTME) Trans-anal Versus Laparoscopic Total Mesorectal Excision for Mid and Low Rectal Cancer
Brief Title: Trans-anal Versus Laparoscopic TME for Mid and Low Rectal Cancer
Acronym: MansTaTME
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammad Zuhdy, Assistant Lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MansTaTME/17.04.84
Record Dates: First submitted 2017-08-01; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Rectal Cancer
Keywords: Minimally invasive surgery; trans-anal total mesorectal excision; Laparoscopic total mesoretal excision
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans-anal TME (TaTME) (Experimental): Trans-anal total mesorectal excision(TaTME) will be offered to patients in this group (assisted by minilaparoscopy to control the IMA and splenic flexure mobilisation)
  Interventions: Procedure: Trans-anal total mesorectal excision(TaTME)
- Lap. TME (Active Comparator): Laparoscopic total mesorectal excision(Lap.TME) starting by IMA ligation then splenic flexure mobilisation and pelvic dissection
  Interventions: Procedure: Lap. TME

INTERVENTIONS:
Procedure: Trans-anal total mesorectal excision(TaTME) — Trans-anal total mesorectal excision(TaTME) will be offered to patients in this group (assisted by minilaparoscopy to control the IMA and splenic flexure mobilisation)
  Other Names: Bottom to up approach
  Arms: Trans-anal TME (TaTME)
Procedure: Lap. TME — Laparoscopic total mesorectal excision(Lap.TME) starting by IMA ligation then splenic flexure mobilisation and pelvic dissection
  Arms: Lap. TME

SUMMARY:
This study is designed to assess the surgical, oncological and functional outcome of either the laparoscopic or trans-anal TME in management of mid and low rectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is considered the third most common type of cancer all over the world and the fourth common cause of cancer-specific mortality.Surgical management for rectal cancer is challenging due to the narrow pelvis and extreme proximity to contiguous organs hence, recurrence rates are commonly reported.

The advent of total mesorectal excision (TME) together with minimally invasive techniques such as laparoscopic colorectal surgery have not only improved surgical results but have also improved surgical technique, operative ability and surgical visibility. Lap TME has been shown to give similar results to the classical open approach with regard to peri-operative morbidity, surgical margins, quality of the surgical specimen, and number of resected lymph nodes, local recurrence and overall survival.

However, laparoscopic resection of mid and low rectal cancer is technically difficult due to tapering of the mesorectum in the pelvis and the forward angle of the distal rectum rendering this part of the rectum less accessible from the abdominal cavity. This may lead to incomplete mesorectal excision and involved circumferential resection margins (CRMs), with consequent local recurrences.Previous pelvic radiation can make laparoscopic pelvic dissection more difficult, and tumors located on the anterior rectal wall have an increased risk of inadequate oncological clearance. The use of laparoscopic staplers in a narrow pelvis is difficult and the multiple firings of staples across the low rectum is of concern.

Trans-anal Total Mesorectal Excision (TaTME) was recently developed to overcome technical difficulties associated with Lap TME and open TME. It may address some of the difficult aspects of laparoscopic or open TME, such as exposure, rectal dissection, and distal cross-stapling of the rectum and sphincter preservation. It does not only facilitate dissection of the difficult distal part of the TME dissection in the narrow pelvis but it also allows clear definition of safe, tumor-free, radial and longitudinal margins. Moreover, the specimen could be extracted through the anus excluding the need for minilaparotmy.

ELIGIBILITY:
Inclusion Criteria:

1. Anesthetically fit patient.
2. Non metastatic pathologically proven rectal cancer (Mid-Low).
3. Patients who received neoadjuvant chemo-radiotherapy will be included

Exclusion Criteria:

1. Patients with American Society of Anesthesiologist (ASA) score 4 and 5.
2. Patients with cardiac or chest problems that cannot withstand CO2 insufflation.
3. Unresectable tumors (T4) (defined as those who cannot be resected without a high likelihood of leaving microscopic or gross residual disease at the local site because of tumor adherence or fixation).
4. Obstructed or perforated cancer.
5. Patients with unresectable metastatic rectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2019-01-25 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Circumferential radial margin (CRM) | 2 years
  Percentage of participants with involved circumferential margin(pathological assessment)
Distal safety margin | 2 years
  Distance of free distal margin in mm (pathological assessment)
Number of lymph nodes retrieved | 2 years
  Number of infiltrated/ Number of harvested lymph nodes(pathological assessment)

SECONDARY OUTCOMES:
Morbidity rate | 2 years
  Number of intra-operative and post-operative encountered complications
Rate of conversion | 2 years
  Percentage of conversion to open technique or to laparoscopy in TaTME cases or open in lap. cases
Disease free survival | 30 months
  Time till development of local or distant recurrence in months
Functional outcome | 18 months
  Assessment of functional outcome via questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Center, Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brenner H, Kloor M, Pox CP. Colorectal cancer. Lancet. 2014 Apr 26;383(9927):1490-1502. doi: 10.1016/S0140-6736(13)61649-9. Epub 2013 Nov 11. PMID 24225001
- [Background] Vennix S, Pelzers L, Bouvy N, Beets GL, Pierie JP, Wiggers T, Breukink S. Laparoscopic versus open total mesorectal excision for rectal cancer. Cochrane Database Syst Rev. 2014 Apr 15;2014(4):CD005200. doi: 10.1002/14651858.CD005200.pub3. PMID 24737031
- [Background] Qu C, Yuan RF, Huang J, Liu L, Jiang CH, Yang ZQ, Shao JH. [Meta-analysis of laparoscopic versus open total mesorectal excision for middle and low rectal cancer]. Zhonghua Wei Chang Wai Ke Za Zhi. 2013 Aug;16(8):748-52. Chinese. PMID 23980046
- [Background] Deijen CL, Velthuis S, Tsai A, Mavroveli S, de Lange-de Klerk ES, Sietses C, Tuynman JB, Lacy AM, Hanna GB, Bonjer HJ. COLOR III: a multicentre randomised clinical trial comparing transanal TME versus laparoscopic TME for mid and low rectal cancer. Surg Endosc. 2016 Aug;30(8):3210-5. doi: 10.1007/s00464-015-4615-x. Epub 2015 Nov 4. PMID 26537907
- [Background] Atallah S, Martin-Perez B, Albert M, deBeche-Adams T, Nassif G, Hunter L, Larach S. Transanal minimally invasive surgery for total mesorectal excision (TAMIS-TME): results and experience with the first 20 patients undergoing curative-intent rectal cancer surgery at a single institution. Tech Coloproctol. 2014 May;18(5):473-80. doi: 10.1007/s10151-013-1095-7. Epub 2013 Nov 23. PMID 24272607
- [Background] Simillis C, Hompes R, Penna M, Rasheed S, Tekkis PP. A systematic review of transanal total mesorectal excision: is this the future of rectal cancer surgery? Colorectal Dis. 2016 Jan;18(1):19-36. doi: 10.1111/codi.13151. PMID 26466751